CLINICAL TRIAL: NCT05529732
Title: The Effect of e-Mobile Education Organized According to Life Model on Anxiety and Daily Living Activities of Patients With Thyroidectomy
Brief Title: The Effect of Mobile Education on Anxiety and Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Muaz Gulsen, Academic Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CukurovaUnıversıty
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Anxiety; Mobile Education; Patient Education; Anxiety; Activities of Daily Living
MeSH Terms: conditions — Anxiety Disorders | interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm randomized controlled clinical trail
Who Masked: Outcomes Assessor
Masking Description: After the researh report is written, a third person will assing an intervention and control group to the letters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Group (Experimental): Oral and written consent will be obtained from the patients by face-to-face interview technique at least one day before the surgery. Then, face-to-face interview technique and data collection tools (Personal Information Form and Trait Anxiety Scale) will be applied. It is estimated that the process of obtaining consent and filling out the form will take approximately 5 minutes. The mobile application will be installed on the mobile devices of the patients and the user name and password will be defined by the researcher so that they can log into the mobile application. In the application, a patient warning notification will be sent on the 3rd, 7th and 10th days to remind the patients to fill in the State Anxiety Scale and Daily Living Activities Evaluation and Follow-up Form, which are included in the questionnaires menu and will be active when the day comes.
  Interventions: Other: e-Mobile Application Patient Education for Patients with Thyroidectomy
- Control Group (No Intervention): Written consent will be obtained from the patients through a face-to-face interview at least one day before the surgery and the data collection form (Personal Information Form and Trait Anxiety Scale) will be filled. During this period, standard care and follow-up protocols will be applied to the patients by the clinic. Patients in the control group will be called by phone on the 3rd, 7th and 10th days of discharge. State Anxiety Scale and Daily Living Activities Evaluation and Follow-up Form will be applied by the researcher. The process is estimated to take 15 minutes.

INTERVENTIONS:
Other: e-Mobile Application Patient Education for Patients with Thyroidectomy — Its mobile application is prepared according to the "Android Operating System" and can be downloaded free of charge from the Google Play Store, it is an application that provides training and consultancy services for patients who have had thyroidectomy surgery.
  Arms: Application Group

SUMMARY:
The study was planned as a block randomized controlled experimental study. In order to calculate the sample size needed in our study, a pilot study will be conducted and a priori power analysis will be made based on the results of this study.

E-mobile application will be used as data collection tool. The research will be carried out with 2 groups as application (mobile application) and control (standard care).

DETAILED DESCRIPTION:
The study was planned as a block randomized controlled experimental study. In order to calculate the sample size needed in our study, a pilot study will be conducted and a priori power analysis will be made based on the results of this study.

E-mobile application will be used as data collection tool. The "E-Mobile Application Training Content Guide" to be integrated into the mobile application will be evaluated by the experts with the "Conformity Evaluation Form of Written Training Materials" and the "DISCERN Scale". After the training content is completed, "Personal Information Form", "STAI State and Trait Anxiety Scale", "Assessment and Monitoring Form for Daily Living Activities" will be used. In the preliminary application, the "System Usability Scale" and the e-mobile application will be evaluated by the patients. The "E-Mobile Application Training Content Guide" created by the researchers in line with the literature will be transferred to the mobile application with the help of computer engineers and graphic designers. Sequence and visuality of education Roper et al. It was designed according to the Life Activities Based Nursing Model developed by The e-mobile application is designed in accordance with the Android operating system and its language is Turkish. Patients who download the application from the virtual market (Google Play) can log in with the user name and password created by the researcher. The user name and password were created by the researcher specifically for each patient during the research process. The number of clicks and the reading time of the topics read by the patients entering the application can be tracked with the help of the created web page. The research will be carried out with 2 groups as application (mobile application) and control (standard care).

ELIGIBILITY:
Inclusion Criteria:

* Thyroidectomy was planned for benign thyroid disease,
* Hospitalized at least one day before the operation,
* Voluntarily accepted to participate in the study,
* Aged 18 and over,
* Conscious, person-space-time orientation,
* No psychiatric problems,
* No hearing-speech and visual impairment
* who can speak Turkish,
* who underwent partial thyroidectomy/lobectomy/total thyroidectomy under general anesthesia and by the same surgeon,
* who have been using a smartphone for at least one year will be included.

Exclusion Criteria:

* Patients with psychiatric problems,
* hearing or speech impairment, who did not approve the informed consent form, who gave up after approval,
* who did not use the mobile application despite using a smartphone,
* who have a profession in the field of health will not be included in the study.
* In addition, patients who did not log into the mobile application, could not be contacted during the research process and whose surgery was canceled for any reason will not be included in the sample.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
STAI State and Trait Anxiety Inventory: | 1 year
  STAI State and Trait Anxiety Inventory: The scale was developed by Spielberger in 1964 and adapted into Turkish by Öner and Le Compte. The scale consists of two parts and includes a total of 40 questions. 20 questions in the first part evaluate the state anxiety of individuals, and 20 questions in the second part evaluate the trait anxiety.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Muaz Gülşen, Adana, Asia
  - Muaz GÜLŞEN, Adana